CLINICAL TRIAL: NCT00710099
Title: Effect of Oral Sildenafil With Digital Therapeutic Iontophoresis of Sodium Nitroprussiate on Cutaneous Blood Flow in Healthy Volunteers
Brief Title: Effect of Oral Sildenafil With Digital Therapeutic Iontophoresis of Sodium Nitroprussiate in Healthy Volunteers
Acronym: INFLUX-VS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCIC/08/08
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: iontophoresis; cutaneous microcirculation; sildenafil; Healthy volunteers
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: sildenafil
- 2 (Active Comparator): SNP iontophoresis
  Interventions: Drug: nitroprussiate iontophoresis

INTERVENTIONS:
Drug: sildenafil — systemic absorption of sildenafil
  Arms: 1
Drug: nitroprussiate iontophoresis — nitroprussiate iontophoresis
  Arms: 2

SUMMARY:
Iontophoresis is a employed to facilitate drug absorption without systemic effect. This study investigates cutaneous microcirculation when we associate sildenafil per os with SNP via iontophoresis.

DETAILED DESCRIPTION:
The main outcome is the proof of concept of effect of systemic absorption sildenafil on cutaneous microcirculation associated with SNP iontophoresis.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* No significant medical history

Exclusion Criteria:

* Age under 18
* Period of exclusion for an other study
* Pregnancy
* Breast feeding
* Severe disease
* Cigarette smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
variation of conductance of nitroprussiate iontophoresis associated with oral sildenafil | one hour

SECONDARY OUTCOMES:
To assess the effect of oral sildenafil (50 mg and 100 mg) on skin microvascular reactivity to local cooling, on the forearm and the finger | one hour

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc CRACOWSKI, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Clinical Researsh Centre, Grenoble, Isere, France

REFERENCES:
- [Background] Cracowski JL, Minson CT, Salvat-Melis M, Halliwill JR. Methodological issues in the assessment of skin microvascular endothelial function in humans. Trends Pharmacol Sci. 2006 Sep;27(9):503-8. doi: 10.1016/j.tips.2006.07.008. Epub 2006 Jul 31. PMID 16876881